CLINICAL TRIAL: NCT05104424
Title: The Study of Quadruple Therapy Intranasal Insulin, Zinc, Gabapentin, Ice Cube Stimulation for Post Covid-19 Smell and Taste Dysfunctions
Acronym: COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Amr kamel khalil Ahmed, clinical researcher and Director of mobile team tuberculosis program, Ministry of Health, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: smell and taste disorders
Record Dates: First submitted 2021-10-25; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Smell Dysfunction; Taste Disorders; Taste Disorder, Secondary, Sweet; Taste Disorder, Secondary, Bitter; Smell Disorder
MeSH Terms: conditions — Olfaction Disorders; Taste Disorders | interventions — Insulin Aspart; Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- adult post covid-19 recovered 22 patients with smell and taste dysfunction take quadruple therapy (Active Comparator): adult patients recovered postcovid-19 taking the quadruple therapy zinc 50 mg , gabapentin 300 mg , 40 I.U rapid insulin , 3 times small cube of ice in the mouth Questionnaires will be administered pre- and post-treatment to assess the change in measures. The mean values between groups will be compared.
  Interventions: Drug: Insulin aspart
- patients taking zinc only with smell training on volatile oils (Placebo Comparator): these 22 adult patients on zinc 50 mg and smell training on 4 volatile oils
  Interventions: Drug: Insulin aspart

INTERVENTIONS:
Drug: Insulin aspart — intranasal rapid insulin 40 I.U as 0.1 ml as 2 puff at each nostril once weekly for 8 weeks zinc 50 mg orally daily Gabapentin 300 mg once daily for 1 month small ice cube at mouth before meals thrice daily
  Other Names: zinc; gabepentin

SUMMARY:
post covid-19 smell and taste dysfunction are common globally and affect the quality of life and also have phycological impact and anxiety, also affect on economy as the patients not able to do cooking or buy prepared foods and not eaten, also not able to enter the cooking room and prepare foods for themselves, also the risk of loss of smell the fire accidents because anosmia, many forms of smell dysfunction like anosmia ,hyposmia, and dysosmia ,Phantosmia , parosmia may occurred, the same taste disorders may has many forms like Dysgeusia, phantom taste perception, hypogeusia with dysgeusia. until now no definite treatments for post covid-19 smell and taste disorders , this study is novel study as quadruple therapy Intranasal Insulin, Zinc, Gabapentin, Ice Cube Stimulation may suspect having promising results

DETAILED DESCRIPTION:
post covid-19 smell and taste dysfunction are common globally and affect the quality of life and also have phycological impact and anxiety, also effect on economy as the patients not able to do cooking or buy prepared foods and not eaten, also not able to enter the cooking room and prepare foods for themselves, also the risk of loss of smell the fire accidents because anosmia, many forms of smell dysfunction like anosmia , hyposmia, and dysosmia , Phantosmia , parosmia may occurred, the same taste disorders may has many forms like Dysgeusia, phantom taste perception, hypogeusia . until now no definite treatments for post covid-19 smell and taste disorders , this study is novel study as quadruple therapy Intranasal Insulin, Zinc, Gabapentin, Ice Cube Stimulation may suspect having promising results.

The application of intranasal insulin in healthy humans has been linked to improve memory function and increased olfactory thresholds also enhance the olfactory performance and regenerate the olfactory epithelium which the corner stone mechanism at affection of smell and taste disorders. zinc orally has many functions and improve taste and influence the activity of carbonic anhydrase in saliva which is important in breaking down foods in our mouth . the application of small ice cube in the mouth for one minute may improve seat taste and lower temperature by 5 degrees. gabapentin working by altering or blocking abnormal electrical discharges arising from the peripheral damaged smell or taste organ

ELIGIBILITY:
Inclusion Criteria:

* adult male or female recovered patients only postcovid-19 no other interventional treatment

Exclusion Criteria:

less than 18 years any nasal deviation or congenital anomalies any allergic sinusitis or nasal problems pregnant women's

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-12-26 (Estimated); Primary Completion 2022-08-26 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of disturbances of smell and taste (Sniffin 'Sticks" test) | 4 month
  The change in smell is based on the comparison of the results of the olfactory assessment after / before treatment obtained from a single method out of the three carried out:
  Sniffin 'Stick Test Results: Threshold Test Score and Actual Identification Test Score.
  TI score: sum of the individual scores of the threshold and identification measures (TI score varying from 0 to 32). It is used to classify patients in terms of normosmia, hyposmia and functional anosmia based on normative values of "Sniffin 'Sticks" (according to the age and sex of each subject) with the threshold at the tenth percentile of the database provided in the study published by Hummel and Kobal.
  Self-assessment by patients using a digital scale of smell, from 0 (no smell) to 10 (normal smell)
evaluation of taste disorders | 4 month
  A device is used to present a pseudo-randomised series of taste solutions to the participant for identification, in order to establish taste thresholds.Change in taste threshold measures (sweet, salt, bitter, sour) between baseline and and post treatment is initiated is assessed with the assistance of a taste test device.
questionnaire for taste self assessment ( Dynachron-olfaction questionnaire) | 4 month
  Self-assessment using the Dynachron-olfaction questionnaire:each question is used to assess the patient's feelings about his discomfort in the nose using a scale from 0 (no discomfort) to 10 (unbearable

SECONDARY OUTCOMES:
any clinical manifestations or adverse effects | 4 month
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0"

IPD SHARING:
Plan to Share IPD: No